CLINICAL TRIAL: NCT00831597
Title: Bendamustine Combined With Rituximab for Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: 904
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmatech (Industry)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI-08904; IND Exemption Number 103985
Record Dates: First submitted 2009-01-26; First posted 2009-01-29 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2012-05

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma; B-Cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine with rituximab (Experimental): All patients received combination bendamustine with rituximab
  Interventions: Drug: bendamustine; Drug: rituximab

INTERVENTIONS:
Drug: bendamustine — 120 mg/m2 IV, Days 1, 2 of Cycles 1-6
  Other Names: Treanda
Drug: rituximab — 375 mg/m2 IV, Day 1 of Cycles 1-6
  Other Names: Rituxan

SUMMARY:
A phase II trial to evaluate the efficacy and safety of combination bendamustine and rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma. It is hypothesized that the BR combination will produce at least a 70% overall response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20-positive, diffuse large B-cell lymphoma
* Measurable disease with at least one bidimensional lymph node or tumor mass > 1.5 cm in the longest diameter that can be followed for response as a target lesion as measured by PET or CT
* Relapsed or refractory after at least one prior therapeutic treatment for diffuse large B-cell lymphoma. Relapsed is defined as patients who initially responded and then progressed. Refractory is defined as patients, whom in the judgment of the Investigator, received adequate prior treatment and did not respond during treatment or progressed within 60 days of last treatment. Relapse following an autologous stem cell transplant allowed.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Patient must understand and voluntarily sign IRB-approved informed consent
* Life expectancy ≥ three (3) months
* Age ≥ 18 years old
* Laboratory parameters:

  * Absolute neutrophil count ≥ 1,000 cells/mm(3)
  * Platelet count ≥ 75,000 cells/mm(3)
  * Hemoglobin ≥ 8 g/dL
  * Creatinine ≤ 2.0 mg/dL or Creatinine Clearance ≥ 50 mL/min (calculated or 24-hr urine sample)
  * AST/SGOT 2.0 x ULN (≤ 5.0 x ULN if secondary to liver metastases)
  * ALT/SGPT 2.0 x ULN (≤ 5.0 x ULN if secondary to liver metastases)
  * Total bilirubin ≤ 2.0 x ULN

Exclusion Criteria:

* Patients with active/symptomatic central nervous system (CNS) involvement based on clinical evaluation. Previously treated CNS involvement that has remained asymptomatic for ≥ 90 days allowed if no CNS involvement shown by lumbar puncture, PET, CT or MRI.
* Prior treatment with bendamustine
* Known sensitivity to bendamustine or any component of bendamustine
* Known anaphylaxis or immunoglobulin E (IgE) mediated hypersensitivity to murine proteins or sensitivity to rituximab or any component of rituximab
* Eligible for stem cell transplant (patients who refuse procedure will not be excluded)
* Prior allogeneic stem cell transplant within 6 months of Cycle 1, Day 1
* Major surgery, not related to debulking procedures, within 21 days of Cycle 1, Day 1. Patients undergoing debulking procedures and minor surgery are allowed after a recovery period, in the judgment of the Investigator.
* Chemotherapy, immunotherapy, or irradiation within 28 days of Cycle 1, Day 1 (within 6 weeks for nitrosoureas or mitomycin). Patients on high dose corticosteroids must have tapered to a stable dose equivalent to Prednisone ≤ 15 mg per day within 28 days of Cycle 1, Day 1.
* Prior radioimmunotherapy (i.e. Zevalin®) within 10 weeks of Cycle 1, Day 1
* Prior use of investigational anti-cancer agents within 28 days of Cycle 1, Day 1
* Unresolved toxicities ≥ grade 2 from previous therapy
* Pregnant or lactating females. Females of childbearing potential (FCBP) and non-vasectomized men must agree to use effective methods of birth control during and 28 days following treatment period. FCBP must have a negative pregnancy test.
* HIV-related lymphoma
* Known active HIV or HCV infection, or known seropositivity for HIV, or current or chronic HBV or HCV infection. HBV test required at screening or within 6 months of screening and must indicate negative result. Patients with seropositivity presumed to be due to prior vaccination against Hepatitis B or resolved infection are not excluded (see HBV reactivation guidelines included in rituximab prescribing information).
* Concurrent active or history of other malignancies, except nonmelanoma skin cancer or carcinoma in situ of cervix or breast. Patients with previous malignancies are eligible provided they have been disease free for ≥ 1 year.
* Serious (grade 3-4), active, intercurrent infection requiring therapy, or deep seated or systemic mycotic infections
* Myocardial infarction within 6 months prior to registration or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or significant conduction system abnormalities, in the judgment of the Investigator
* Thyroid disease in which thyroid function cannot be maintained within normal range, in the judgment of the Investigator
* Concurrent uncontrolled serious medical or psychiatric conditions likely to interfere with participation in this clinical study, in the judgment of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Best Overall Response Rate (ORR) of bendamustine in combination with rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma | 1 year for 1st assessment and then 2.5 years for final assessment

SECONDARY OUTCOMES:
Duration of Response (DOR) | 1 year for 1st assessment and then 2.5 years for final assessment
Time to Progression (TTP) | 1 year for 1st assessment and then 2.5 years for final assessment
Progression-Free Survival (PFS) | 1 year for 1st assessment and then 2.5 years for final assessment
Safety Profile of Study Treatment | 1 year for 1st assessment and then 2.5 years for final assessment
Overall Survival (OS) | 1 year for 1st assessment and then 2.5 years for final assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Vacirca, MD, FACP, Principal Investigator — University Hospital, Stony Brook North Shore Hematology/Oncology Associates
Locations (32):
- United States (32):
  - Pharmatech Oncology Study Site, Beverly Hills, California
  - Pharmatech Oncology Study Site, Fountain Valley, California
  - Pharmatech Oncology Study Site, Oxnard, California
  - Pharmatech Oncology Study Site, Washington D.C., District of Columbia
  - Pharmatech Oncology Study Site, Boynton Beach, Florida
  - Pharmatech Oncology Study Site, Brooksville, Florida
  - Pharmatech Oncology Study Site, Gainesville, Florida
  - Pharmatech Oncology Study Site, Titusville, Florida
  - Pharmatech Oncology Study Site, Joliet, Illinois
  - Pharmatech Oncology Study Site, Lafayette, Indiana
  - Pharmatech Oncology Study Site, Muncie, Indiana
  - Pharmatech Oncology Study Site, Dubuque, Iowa
  - Pharmatech Oncology Study Site, Paducah, Kentucky
  - Pharmatech Oncology Study Site, York Village, Maine
  - Pharmatech Oncology Study Site, Jackson, Mississippi
  - Pharmatech Oncology Study Site, Chesterfield, Missouri
  - Pharmatech Oncology Study Site, Cherry Hill, New Jersey
  - Pharmatech Oncology Study Site, Phillipsburg, New Jersey
  - Pharmatech Oncology Study Site, Bay Shore, New York
  - Pharmatech Oncology Study Site, East Setauket, New York
  - Pharmatech Oncology Study Site, The Bronx, New York
  - Pharmatech Oncology Study Site, Akron, Ohio
  - Pharmatech Oncology Study Site, Columbus, Ohio
  - Pharmatech Oncology Study Site, Bethlehem, Pennsylvania
  - Pharmatech Oncology Study Site, Gettysburg, Pennsylvania
  - Pharmatech Oncology Study Site, Hilton Head, South Carolina
  - Pharmatech Oncology Study Site, Germantown, Tennessee
  - Pharmatech Oncology Study Site, Austin, Texas
  - Pharmatech Oncology Study Site, Corpus Christi, Texas
  - Pharmatech Oncology Study Site, Fort Worth, Texas
  - Pharmatech Oncology Study Site, Lubbock, Texas
  - Pharmatech Oncology Study Site, Richardson, Texas

REFERENCES:
- [Result] Vacirca JL, Acs PI, Tabbara IA, Rosen PJ, Lee P, Lynam E. Bendamustine combined with rituximab for patients with relapsed or refractory diffuse large B cell lymphoma. Ann Hematol. 2014 Mar;93(3):403-9. doi: 10.1007/s00277-013-1879-x. Epub 2013 Aug 17. PMID 23955074
- See also: Related Info — http://www.pharmatech.com
- See also: Related Info — http://abstract.asco.org/AbstView_74_51249.html
- See also: Study Publication Abstract — http://www.ncbi.nlm.nih.gov/pubmed/23955074